CLINICAL TRIAL: NCT04631211
Title: A Prospective, Multicenter, Randomized, Open-Label Phase 2, Parallel, Dose Ranging Multidose Study of Thrombosomes® vs Liquid Stored Platelets (LSP) in Bleeding Thrombocytopenic Patients
Brief Title: Thrombosomes® in Bleeding Thrombocytopenic Patients Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to loss of funding for this indication from the Biomedical Advanced Research and Development Authority (BARDA) in November 2022.
Sponsor: Cellphire Therapeutics, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #2019-1
Expanded Access: NCT04619108 (No longer available)
Record Dates: First submitted 2020-11-05; First posted 2020-11-17 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Thrombocytopenia; Hematologic Malignancy; Bone Marrow Aplasia; Myeloproliferative Disorders; Myelodysplastic Syndromes; Platelet Refractoriness
MeSH Terms: conditions — Thrombocytopenia; Hematologic Neoplasms; Anemia, Aplastic; Myeloproliferative Disorders; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: Dose Ranging Multidose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Thrombosomes Low Dose (Experimental)
  Interventions: Biological: Thrombosomes
- Thrombosomes Medium Dose (Experimental)
  Interventions: Biological: Thrombosomes
- Thrombosomes High Dose (Experimental)
  Interventions: Biological: Thrombosomes
- Liquid Stored Platelets (Control) (Active Comparator)
  Interventions: Biological: Liquid Stored Platelets (LSP)

INTERVENTIONS:
Biological: Thrombosomes — Human platelet derived lyophilized hemostatic
  Arms: Thrombosomes High Dose; Thrombosomes Low Dose; Thrombosomes Medium Dose
Biological: Liquid Stored Platelets (LSP) — Leukocyte reduced apheresis platelets or whole blood derived pooled platelet concentrate equivalent (4-6 units)
  Arms: Liquid Stored Platelets (Control)

SUMMARY:
This prospective, multicenter, randomized, open-label, Phase 2, parallel, dose ranging, multidose trial will enroll patients into 3 Thrombosomes dose groups and 1 control liquid stored platelets (LSP) group in order to evaluate, in a dose-escalation manner, the safety, and impact on bleeding, and the preliminary effect on coagulation measures of increasing doses of allogeneic Thrombosomes in comparison to standard of care, LSP.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) with TCP as defined by BOTH (a) and (b):

   1. a platlet count of ≤ 70,000 platelets/μL blood
   2. ANY ONE OR MORE of (1-3):

      1. confirmed diagnosis of hematologic malignancy, myeloproliferative disorder, myelodysplastic syndrome, or aplasia
      2. undergoing chemotherapy, immunotherapy, radiation therapy or hematopoietic stem cell transplantation
      3. refractory to platelet transfusion defined as two 1-hour CCI of <5,000 on consecutive transfusions of LSP or as defined by local site policy (Sacher, 2003)
2. WHO Bleeding Score of 2 or 3
3. Able to provide informed consent directly or through legally authorized representative, and comply with treatment and monitoring
4. Negative pregnancy test for women of childbearing potential

Exclusion Criteria:

1. Any disorder or condition related to any venous thrombosis, embolism, or ischemia within the past 3 months
2. Any disorder or condition related to arterial thrombosis including: ischemia, stroke, MI, or stent placement, within past 6 months
3. Any valve replacement and/or repair of left atrial appendance occlusion device
4. Sinusoidal obstruction syndrom (veno-occlusive disease) or cytopkine release syndrome associated with CAR-T cell therapy
5. Refusal to accept blood products
6. Liver enzyme blood levels greater than 3× the upper limit of normal (ULN)
7. Blood creatinine level greater than 3× ULN
8. Received platelet inhibitor drugs, cyclooxygenase-2 (COX-2) inhibitors, or nonsteroidal anti-inflammatory drugs within 5 days prior to infusion
9. Currently (at the time of randomization) receiving anticoagulant therapy or antiplatelet therapy. Low dose prophylaxis for line clots is not excluded.
10. Receipt of any pro-coagulant agents (e.g., DDAVP, recombinant Factor VIIa or prothrombin complex concentrates (PCC)) other than Tranexamic Acid (TXA) or Epsilon Aminocaproic Acid (EACA, Amicar), within 48 hours of first infusion, or with known hypercoagulable state
11. WHO Bleeding Score of 2 solely due to lumbar puncture, retinal bleeding or GI bleeding or WHO Bleeding Score of 3 solely due to lumbar puncture
12. Receiving L-asparaginase as part of a current cycle of treatment
13. Known inherited or acquired bleeding disorder including, but not limited to: acquired storage pool deficiency or paraproteinemia with platelet inhibition
14. Known inherited or acquired prothrombotic disorders, including antiphospholipid syndrome (Those with lupus anticoagulant or positive antiphospholipid serology without thrombosis are NOT excluded.)
15. Anuria
16. On dialysis
17. Receipt of an investigational drug within 1 month before first infusion, other than for treatment of their underlying disease
18. Females pregnant or nursing or unwilling to use contraception during and for 30 days after taking the study product (females). Evidence of effective birth control may be used, at the discretion of the physician
19. Acute or chronic medical disorder that, in the opinion of the Investigator, would impair the ability of the patient to receive or respond to study treatment
20. Prior participation in this study with successful infusion of the investigational or control product
21. Currently enrolled in other trials not related to their primary disease process or involving platelet transfusions, platelet growth factors, or other pro-coagulant agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | Evaluated at 24 hours post initial infusion
  Cessation or decrease in bleeding at primary bleeding site, based upon the most severe bleeding location at Day 1 baseline taken with in 12 hours prior to infusion, as evidenced by ordinal change in WHO (World Health Organization) Bleeding Score evaluated at 24 hours post initial infusion.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint assessed by Number of days alive and without WHO (World Health Organization) Grade 2a or greater bleeding | 7 days after first Thrombosomes or LSP infusion
  Number of days alive and without WHO (World Health Organization) Grade 2 or greater bleeding through initial 7 days after first Thrombosomes or LSP Infusion
Secondary Efficacy Endpoint assessed by 30 day mortality | 30 days post first infusion (+/- 2 days)
  30-day mortality post first infusion of Thrombosomes or post first infusion of LSP as control
Secondary Efficacy Endpoint assessed by cessation or decrease in bleeding, as evidenced by ordinal change in WHO (World Health Organization) Bleeding Score | 24, 48, 72 hours, Day 4, Day 5, Day 6 and Day 7 post first infusion
  Cessation or decrease in primary bleeding site, as evidenced by ordinal change in WHO (World Health Organization) Bleeding Score at 24, 48, 72 hours, Day 4, Day 5, Day 6 and Day 7 after first infusion of Thrombosomes or LSP infusion as control.
Secondary Efficacy Endpoint assessed by cessation or decrease in bleeding, as evidenced by ordinal change in WHO (World Health Organization) Bleeding Score | 24, 48, 72 hours, Day 4, Day 5, Day 6 and Day 7 post first infusion
  Cessation or decrease in each additional bleeding site (other than primary bleeding site), as evidenced by ordinal change in WHO (World Health Organization) Bleeding Score at 24, 48, 72 hours, Day 4, Day 5, Day 6 and Day 7 after first infusion of Thrombosomes or LSP infusion as control.
Secondary Efficacy Endpoint assessed for Number, timing, type and reason for administration of all blood products | 7 days after first Thrombosomes or LSP infusion
  Number, timing, type and reason for administration of all blood products including platelets and Thrombosomes during the initial 7 days after first Thrombosomes or LSP infusion
Secondary Efficacy Endpoint assessed by platelet count | 24, 48, 72 hours and Day 7 post first infusion
  Platelet count measured at 24, 48, 72 hours and Day 7 of first infusion of Thrombosomes or LSP. Also evaluate at Day 4-6 if patient is hospitalized at that time.
Secondary Efficacy Endpoint assessed by measures of hematology | From baseline through last study visit (up to 30 days (+/- 2 days))
  Measures of hematology including: Prothrombin Fragment 1+2; thrombin generation assay (TGA); Thrombopoietin; activated Protein C, tissue plasminogen activator (TPA), and plasminogen activator inhibitor (PAI) per schedule of assessments
Secondary Efficacy Endpoint assessed by measures of coagulation | From baseline through last study visit (up to 30 days (+/- 2 days))
  Measures of coagulation including: prothrombin time (PT); international normalized ratio (INR); fibrinogen; D-dimer; activated partial thromboplastin time (aPTT); and thromboelastography (TEG) or rotational thromboelastometry (ROTEM) per schedule of assessments
Secondary Efficacy Endpoint assessed by changes in markers of endothelial cell injury/repair | From baseline through last study visit (up to 30 days (+/- 2 days))
  Changes in markers of endothelial cell injury/repair from preinfusion baseline through 72 hours after first infusion, including: Syndecan-1, hyaluronan, thrombomodulin, vascular endothelial growth factor (VEGF), interleukin 6, sVE cadherin per schedule of assessments.

OTHER OUTCOMES:
Safety Endpoint | From baseline through last study visit (up to 30 days (+/- 2 days))
  Serious Adverse Events (SAEs)
Safety Endpoint | From baseline through last study visit (up to 30 days (+/- 2 days))
  Adverse Events (AEs)
Safety Endpoint | From baseline through last study visit (up to 30 days (+/- 2 days))
  Unanticipated problems involving risk to human subjects

CONTACTS AND LOCATIONS:
Overall Officials: Terry Gernsheimer, MD, Principal Investigator — University of Washington; Mike Fitzpatrick, PhD, Study Director — Cellphire Therapeutics, Inc.
Locations (6):
- United States (4):
  - City of Hope, Duarte, California
  - Medstar Georgetown, Washington D.C., District of Columbia
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Rambam Medical Center, Haifa, Israel
- Helse Bergen Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04631211/ICF_000.pdf